CLINICAL TRIAL: NCT00623168
Title: A Phase 2 Treatment Protocol of Intravenous Ribavirin in Adult Subjects With Hemorrhagic Fever With Renal Syndrome (HFRS) in the 121st Combat Support Hospital (Seoul, Korea)
Brief Title: Ribavirin for Hemorrhagic Fever With Renal Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This was an expanded access treatment protocol that did not enroll any subjects due to no infections requiring treatment.
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-14474; TAMC HUC 23H07 (Other: IRB)
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Hemorrhagic Fever With Renal Syndrome
Keywords: Ribavirin; Hemorrhagic Fever with Renal Syndrome
MeSH Terms: conditions — Hemorrhagic Fever with Renal Syndrome | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Only (Experimental): All consented subjects who meet all inclusion and no exclusion criteria will enter this open label protocol and be treated with Ribavirin.
  Interventions: Drug: Ribavirin

INTERVENTIONS:
Drug: Ribavirin — 7 Day multiple dosing regime based on weight and dosage day

SUMMARY:
Hemorrhagic Fever with Renal Syndrome (HFRS) is caused by a virus acquired by contact with chronically infected rodent hosts. HFRS is present throughout Korea. Treatment consists mainly of supportive care with careful attention to control of blood pressure and fluid balance and/or dialysis. Early initiation of IND Intravenous Ribavirin has been shown to be an effective treatment for HFRS and may prevent the need for dialysis. It is important to initiate therapy based on a diagnosis consistent with HFRS and a history that makes exposure likely. This study will monitor the clinical events that occur with HFRS as well as the safety and efficacy of Ribavirin.

DETAILED DESCRIPTION:
Hemorrhagic Fever with Renal Syndrome (HFRS) is caused by viruses in the genus Hantavirus of the family Bunyaviridae. There are four known Hantavirus that cause HFRS: Hantaan, Seoul, Puumala and Dobrava viruses. HFRS is acquired by contact with chronically infected rodent hosts, most commonly from inhalation of infected rodent excreta. Hemorrhagic fever with renal syndrome is characterized clinically by the triad of fever, hemorrhage and renal insufficiency. HFRS typically consists of five consecutive but frequently overlapping clinical phases: febrile, hypotensive, oliguric, diuretic and convalescent. DoD operations have resulted in the deployment of personnel in Europe and Southeast Asia, areas endemic for HFRS, a viral hemorrhagic fever. Early initiation of therapy with intravenous Ribavirin has been shown to be an effective treatment for HFRS. It is therefore important to initiate therapy based on a clinical diagnosis consistent with viral hemorrhagic fever and with an epidemiological history for risk of exposure to the hantavirus. Ribavirin is a nucleoside (guanosine) analog with activity against a wide variety ribonucleic acid and deoxyribonucleic acid viruses. Mechanism of action is not fully defined. The mechanism may be related to alteration of cellular nucleotide pools and of viral messenger RNA formation, but recent data suggest the mechanism of Ribavirin in HFRS may be to serve as a RNA virus mutagen resulting in an "extinction catastrophe" error, as a result of incorporation in the viral RNA genome.

Ribavirin is licensed in the United States in aerosol form for the treatment of severe lower respiratory tract infection in children and in the oral formulation in combination with recombinant interferon alpha for the treatment of chronic hepatitis C infection. The intravenous formulation of ribavirin in not licensed in the United States. IV Ribavirin for the treatment of HFRS is used under IND 16,666.

This is a Phase 2, open-label study of the safety of IV Ribavirin treatment in individuals with Hemorrhagic Fever with Renal Syndrome (HFRS) admitted to the 121st Combat Support Hospital, Seoul, Republic of Korea. The study will also monitor morbidity and mortality of subjects with HFRS who are treated with IV Ribavirin. The study population will include all subjects with a probable or suspected clinical diagnosis of HFRS, at least 18 years of age (age 17 if active military) but not greater than 65 years of age. The Investigators intend to treat all individuals who present with a tentative diagnosis of HFRS (and within 7 days of onset of illness) and meet entry criteria with a 7 day course of IV Ribavirin and a 28-60 day follow up period after first dose of Ribavirin. In addition to treatment with Ribavirin, all subjects will be given standard supportive and symptomatic care as determined by the clinical judgment of attending physicians or consultants who manage the subject's care at the 121 CSH. Up to 50 subjects could potentially be enrolled in a five year time period with an expected accrual of 0-5 subjects per year, but the number may be higher (10 to 20 persons in a year) if an HFRS outbreak should occur. Specific inclusion/exclusion/relative exclusion criteria are a part of the protocol. Safety procedures required during 7 days of treatment include continuous cardiac monitoring, daily lab work, physical exams and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Have read and signed the Informed Consent (see Exception for Emergency Treatment, Section 12.0).
* Are at least 18 years of age (17, if active military) and not greater than 65 years of age.
* Meet the case definition for a probable or suspected case (see Section 5.0).
* Have a blood sample drawn and a type and cross-match ordered for transfusion.
* Agree to collection of required specimens.
* Agree to report any Adverse Events, Serious and Unexpected Adverse Events for the duration of the study.
* Agree to a follow-up visit and to donate blood and urine specimens at day 10, day 14 and between days 28 and 60 after the first dose of IV Ribavirin and to all follow-up visits for anemia or other medical conditions as required by the attending physician.
* Women of childbearing age must have a negative pregnancy test and agree not to become pregnant for 7 months after receiving Ribavirin. Women will be counseled concerning the risks of IV Ribavirin.
* Men agree not to have intercourse with pregnant women for 7 months after receiving Ribavirin, and take precautions to avoid producing pregnancies for 7 months after receiving Ribavirin.
* Have a hemoglobin greater than or equal to10 g/dL before starting IV Ribavirin.

Exclusion Criteria:

* A known intolerance to Ribavirin.
* Are irreversibly ill on presentation, as defined by presence of profound shock, which does not respond to supportive therapy within 3 hours after admission.
* A positive pregnancy test.
* An estimated creatinine clearance < 20 ml/minute.
* A history of hemoglobinopathies (i.e., sickle-cell anemia or thalassemia major).
* A history of autoimmune hepatitis.
* A hemoglobin less than 10 g/dL that cannot be corrected to ≥10 g/dL before initiation of IV Ribavirin.
* A New York Heart Association Cardiac functional capacity of Class II or greater for ASHD and CHF.
* Known cardiac conduction defects that may predispose the subject to arrhythmias, such as second or third degree heart block or sick sinus syndrome (and no pacemaker), or Wolfe-Parkinson-White Syndrome.
* A sinus bradycardia of less than 40 beats per minute (or sinus bradycardia less than 50 beats per minute if the individual is not known to have a low resting heart rate related to physical conditioning).
* Concurrent therapy with Didanosine (ddI). DdI must be discontinued before starting the IV Ribavirin.

Relative Exclusion Criteria: PI's discretion to use IND Ribavirin with caution. The PI should make the decision concerning enrollment of subjects with relative exclusion criteria based on risk versus benefit of the drug.

* Creatinine clearance is 20 - 30 mL/minute
* History of gout or tophaceous gout
* On any drug that may decrease heart rate (beta-blockers, calcium channel blockers, digoxin IV Ribavirin should be avoided in severe renal insufficiency, and its use with a creatinine clearance between 20 to 30 mL/min should be based on the risk versus benefit. If used, the drug should be discontinued if the creatinine clearance decreases to 20 mL/min or lower.

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Number clinical events that occur with HFRS including oliguria, dialysis requirement, cardiac arrhythmias, and severe hemorrhage | 5 years
Number of mortalities | 5 years

SECONDARY OUTCOMES:
Number and nature of adverse events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Cashin, DO, Principal Investigator — Brian Allgood Army Community Hospital (121st Combat Support), Seoul, Republic of Korea
Locations (1):
- Brian Allgood Army Community Hospital (121st Combat Support), Seoul, South Korea